CLINICAL TRIAL: NCT00641602
Title: A Multicenter, Randomized, Double Blind, Double Dummy, Parallel-Group Efficacy Study Comparing 8 Weeks of Treatment With Esomeprazole Magnesium (40mg qd) to Lansoprazole (30mg qd) for the Healing of Erosive Esophagitis in Patients With Moderate or Severe Erosive Esophagitis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, Astra Zeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 322; D9612L00046
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Erosive Esophagitis
Keywords: Erosive Esophagitis; Nexium; Heartburn
MeSH Terms: conditions — Heartburn | interventions — Esomeprazole; Lansoprazole

ARMS (2):
- 1 (Experimental): Nexium
  Interventions: Drug: Esomeprazole
- 2 (Active Comparator): Prevacid
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Esomeprazole — 40mg once daily
  Other Names: Nexium
  Arms: 1
Drug: Lansoprazole — 30mg once daily
  Other Names: Prevacid
  Arms: 2

SUMMARY:
This study looks at the healing rates in patients with Erosive Esophagitis (EE) when treated with either esomeprazole or lansoprazole

ELIGIBILITY:
Inclusion Criteria:

* Episodes of heartburn (described as a burning feeling, rising from the stomach or lower part of the chest up towards the neck) for 2 days or more during the last 7 days prior to baseline.
* Confirmed Erosive Esophagitis within 1 week prior to starting the study.

Exclusion Criteria:

* Any signs of gastrointestinal bleeding at the time of the starting the study.
* Any previous gastric or esophageal surgery.
* Various gastrointestinal diseases as listed in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2002-12; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
To compare the difference in healing rates of erosive esophagitis (EE) between esomeprazole 40 mg qd (E40) and lansoprazole 30 mg qd (L30) in patients with moderate or severe EE, defined as Grade C or D in the Los Angeles (LA) Classification scale. | Esophagogastroduodenoscopy (EGD) at baseline and then week 4 and week 8 (if not healed at week 4)

SECONDARY OUTCOMES:
1. To compare the difference in the resolution of, and relief of, the investigator evaluated GERD symptoms of heartburn, acid regurgitation, dysphagia, and epigastric pain between E40 and L30 at week 4 of treatment in patients with moderate or severe EE. | Esophagogastroduodenoscopy (EGD) at baseline and then week 4 and week 8 (if not healed at week 4)
1. To compare the difference between E40 and L30 in the occurrence of heartburn symptoms as reported in the patient's daily diary. | Dairy card to be completed by patient daily
To evaluate safety and tolerability of E40 compared to that of L30 in patients with moderate or severe EE. | Adverse event collection on an ongoing basis

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca